CLINICAL TRIAL: NCT00450138
Title: An Open Label Phase 1 Study to Assess the Maximum Tolerated Dose of ZACTIMA™ Given Concomitantly With Weekly Cisplatin Chemotherapy and Radiation Therapy in Patients With Previously Untreated, Unresected Stage III-IV Head and Neck Squamous Cell Carcinoma
Brief Title: Open Label, Phase I ZD6474 Head and Neck Cancer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00062; NCT00411710 (obsolete NCT alias)
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — vandetanib; Cisplatin; Radiation

ARMS (2):
- 1 (Experimental): Radiation + vandetanib
  Interventions: Drug: ZD6474 (vandetanib); Radiation: Radiation
- 2 (Experimental): Radiation + cisplatin + vandetanib
  Interventions: Drug: ZD6474 (vandetanib); Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: ZD6474 (vandetanib) — once daily oral dose
  Other Names: ZACTIMA™
Drug: Cisplatin — intravenous infusion
  Arms: 2
Radiation: Radiation — radiation of head and neck

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of ZD6474 given in combination with radiation or in combination with chemotherapy and radiation in patients with squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Stage III-IV squamous cell carcinoma of the head and neck

Exclusion Criteria:

* No previous treatment for head and neck cancer, adequate cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-12; Primary Completion 2009-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of vandetanib given in combination with radiation or radiation and chemotherapy in patients with late stage head and neck cancer | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Research Site, Denver, Colorado
  - Research Site, Chicago, Illinois
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas

REFERENCES:
- See also: CSR-D4200C00062.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1431&filename=CSR-D4200C00062.pdf
- See also: protocol redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1431&filename=D4200C00062_Clinical_study_revised_protocol_redacted_[SECURE].pdf